CLINICAL TRIAL: NCT04917731
Title: Botulinum Toxin Type A for Cold Intolerance Secondary to Digital Amputations and Replantations: A Pilot Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Jonathan M. Winograd, M.D., Visiting Surgeon, Associate Professor Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002873
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Cold Intolerance
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox (Experimental): The patients in this arm will receive Botox injection to the digital arteries of all affected digits.
  Interventions: Drug: Botulinum toxin type A
- Placebo (Placebo Comparator): The patients in this arm will receive placebo injection of saline to the digital arteries of all affected digits.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Botox injected at digital artery
  Other Names: Botox

SUMMARY:
Patients will be selected for cold intolerance after finger amputation or replantation. They will be given Botox or placebo dose as treatment and assessed over 3 months.

DETAILED DESCRIPTION:
Aim 1: To assess the efficacy of botulinum toxin type A on treating cold intolerance secondary to digital amputations, revascularizations, or replantations

Primary null hypothesis: Randomized subjects who receive botulinum toxin type A injections for pain associated with cold intolerance will experience similar changes in pain as compared to patients randomized to receive saline injections (control)

• As measured by the Cold Insensitivity and Severity Score (CISS) at one week, four weeks, and twelve weeks

Aim 2: To assess the safety of botulinum toxin type A on treating cold intolerance secondary to digital amputations and replantations

Hypothesis: Injection of botulinum toxin for cold intolerance secondary to digital amputations and replantations is not associated with any adverse reactions

III. SUBJECT SELECTION All adult, English-speaking patients who present with cold intolerance secondary to digital amputation or replantation will be approached and asked to participate in the study.

Inclusion criteria Adults (≥18 years) diagnosed with cold intolerance secondary to digital amputations, revascularizations, or replantations and a CISS score of 30 or higher (the threshold for pathological cold intolerance)11 Ability to give informed consent

Exclusion criteria Adults ≥ 75 years old Inability or unwillingness to participate in CISS or DASH survey Major medical comorbidity expected to worsen in the next 6 months Comorbid chronic pain condition Severe and untreated mental health conditions or active substance dependence Pregnant or breastfeeding Known hypersensitivity to botulinum toxin Patients with a compromised respiratory function Pre-existing neuromuscular disorders Receiving therapy with aminoglycosides, anticholinergic agents, and muscle relaxants Infection in the proposed injection site

All patients who satisfy the inclusion/exclusion criteria will be eligible for enrollment. Vulnerable populations will be excluded from this study.

IV. SUBJECT ENROLLMENT A total of twenty-eight patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with cold intolerance secondary to digital amputations, revascularizations, or replantations and a CISS score of 30 or higher (the threshold for pathological cold intolerance)11 Ability to give informed consent

Exclusion Criteria:

* Adults ≥ 75 years old Inability or unwillingness to participate in CISS or DASH survey Major medical comorbidity expected to worsen in the next 6 months Comorbid chronic pain condition Severe and untreated mental health conditions or active substance dependence Pregnant or breastfeeding Known hypersensitivity to botulinum toxin Patients with a compromised respiratory function Pre-existing neuromuscular disorders Receiving therapy with aminoglycosides, anticholinergic agents, and muscle relaxants Infection in the proposed injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-06-02 (Estimated); Study Completion 2023-06-02 (Estimated)

PRIMARY OUTCOMES:
Cold Intolerance Severity Score | 3 months
  index of cold intolerance, validated
quick dash | three months.
  a validated measure of hand function

SECONDARY OUTCOMES:
PHQ 9 | 3 months
  depression measure, validated

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Winograd, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No